CLINICAL TRIAL: NCT02766985
Title: Rasch-analysis of Clinical Severity in FSHD
Acronym: ROC-FSHD
Status: Completed | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: STUDY00003640; UL1TR000001 (NIH)
Record Dates: First submitted 2016-03-22; First posted 2016-05-10 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Facioscapulohumeral Muscular Dystrophy
Keywords: FSHD; muscular dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Facioscapulohumeral; Muscular Dystrophies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples will be collected and stored for genetic testing. Muscle biopsies are also being collected for future functional assays to verify identified genetic modifiers.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- FSHD: Participants with FSHD-1 or FSHD-2. No intervention is given to participants. Participants will undergo series of tests and procedures in order to make a standardized and scalable Rasch-built clinical severity scale.

SUMMARY:
The purpose of this study is to make a standardized and scalable Rasch-built clinical severity scale to help in finding genetic and environmental modifiers of disease in Facioscapulohumeral muscular dystrophy (FSHD).

ELIGIBILITY:
Inclusion Criteria:

* Genetic confirmation of FSHD (either FSHD-1 or FSHD-2)

Exclusion Criteria:

* Do not understand English
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Particpants with genetically verified FSHD types 1 and 2.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2016-03; Primary Completion 2017-04-18 (Actual); Study Completion 2017-04-18 (Actual)

PRIMARY OUTCOMES:
FSHD Clinical Severity Scale | 1 day
  Measure severity of FSHD.

SECONDARY OUTCOMES:
Brooks scale | 1 day
  Measures upper extremity function.Scores on the scale range from 1-6. A score of 1 means the person can elevate their arms above their head while arms remain straight. 6 means the person cannot elevate their arms to their mouth and do not have useful function of their hands.
Vignos scale | 1 day
  Measures lower extremity function. Scores on the scale range from 1-10. A score of 1 means the person can walk and climb stairs without assistance. A score of 10 means the person is bedridden.
Iowa Oral Performance Instrument (IOPI) | 1 day
  IOPI measures lip and tongue strength by measuring the amount of pressure a person can exert on the tool.
Manual muscle testing | 1 day
  Measure person's range of motion. Scored on a scale with range of 0-5. Score of 0 means no movement. Score of 5 means the person has a full range of movement.
Quantitative strength testing | 1 day
Functional testing | 1 day
Reparatory function testing | 1 day
Patient-reported outcome | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Statland, MD, Principal Investigator — University of Kansas Medical Center
Locations (2):
- United States (2):
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Utah, Salt Lake City, Utah